CLINICAL TRIAL: NCT00181675
Title: A Double-Blind Comparison of Galantamine HBr and Placebo in Adults With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Joseph Biederman, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2002-P-001937
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: ADHD
Keywords: Adult; ADHD; galantamine; double-blind
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Galantamine

INTERVENTIONS:
Drug: galantamine HBr

SUMMARY:
This will be a double-blind, placebo-controlled, study using daily doses of up to 24 mg/ day Galantamine HBr in the treatment of adults who meet DSM-IV criteria for childhood-onset ADHD. Specific hypotheses are as follows:

Hypothesis 1: ADHD symptomatology in adults with DSM-IV ADHD will be responsive to acute Galantamine HBr treatment.

Hypothesis 2: Galantamine HBr -associated improvement in ADHD symptomatology in adults will translate into improved functional capacities (neuropsychological, social, and occupational) as well as an increased quality of life throughout acute treatment.

Hypothesis 3: Galantamine HBr treatment will be safe and well tolerated as reflected by a low drop out rate and absence of major differences from placebo.

DETAILED DESCRIPTION:
Galantamine HBr, a tertiary alkaloid, is a competitive and reversible inhibitor of acetylcholinesterase that is indicated to slow the deterioration of cognitive impairment in Alzheimer's Disease. Initial anecdotal data suggest a promising role for Galantamine HBr in the treatment of ADHD. We propose to study to test the safety and efficacy of Galantamine HBr therapy in adults with ADHD. We will test if Galantamine HBr -associated improvements in ADHD symptomatology translate into improved cognitive and functional capacities (social and occupational) as well as increased quality of life.

The proposed study includes 1) use of a 12-week design to document the response rate 2) assessment of the impact of Galantamine HBr on functional capacities (quality of life, psychosocial function) and cognition, 3) careful assessment of safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Male outpatients between 18 to 58 years of age (inclusive).
2. Females between 18 to 58 years of age (inclusive) that are on reliable and adequate birth control.
3. Subjects with the DSM-IV diagnosis of childhood onset Attention-Deficit/Hyperactivity Disorder (ADHD), as manifested in the clinical evaluation and confirmed by structured interview.
4. Subjects with a score of 24 or greater on the ADHD Rating Scale.

Exclusion Criteria:

1. Any current, non-ADHD Axis I psychiatric condition of clinical significance.
2. Baseline Ham-D > 16, BDI > 19, and/or Ham-A > 21.
3. Any clinically significant chronic medical condition, specifically cardiovascular, gastrointestinal, pulmonary, genitourinary, metabolic, or endocrine disorders, and hepatic or renal impairment.
4. Clinically significant abnormal baseline laboratory values.
5. I.Q. <75.
6. Organic brain disorders.
7. Subjects with a history of or current seizure disorders.
8. Pregnant and/or nursing females.
9. Clinically unstable psychiatric conditions (i.e. suicidal behaviors, psychosis).
10. Subjects currently (within the past 6 months) known to abuse or to be dependent on any drug, including alcohol.
11. Subjects on other psychotropic medications, with the exception of SSRIs.
12. Subjects with a history of intolerance or non-response to cholinergic agents as determined by the clinician.
13. Subjects with a history of peptic ulcer disease, gastroesophageal reflux disease, or other GI disorders.
14. Subjects with history of bradyarrythmias.
15. Subjects with asthma.
16. Subjects on ketoconazole.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40
Dates: Start 2002-12; Study Completion 2003-09

PRIMARY OUTCOMES:
symptom reduction using ADHD- Clinical Global Impression & ADHD Symptom Checklist Severity Scale administered weekly

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States